CLINICAL TRIAL: NCT03730272
Title: The Incidence and Strenght of Pain in Conscious Multitrauma Patients, 0-14 Days After Multitrauma
Brief Title: Occurence of Pain and Use of Analgesic Treatment in Multi-trauma Patients of Intermediate Seveity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Johan C Ræder, professor, Oslo University Hospital
Other Study IDs: Trauma.pain.Gyda
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Post Traumatic Pain; Post Traumatic Analgesic Treatment
MeSH Terms: interventions — Analgesics; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: analgesic drugs and methods — the patient will receive analgesic treatment at the discretion of the physician in charge

SUMMARY:
To register the perceived pain score during 0-14 days after multitrauma in conscious patients and to register the use (type and dose) of analgesic treatment in the same period.

ELIGIBILITY:
Inclusion Criteria:

* Patient With trauma, ISS > 8

Exclusion Criteria:

* Unconscious patients at admission
* patients due for major surgery within 3 hrs of admission
* patients primary admitted to other hospitals
* not able to communicate in Norewegian

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients With any kind of multitrauma, fullfilling inclusion/exclusion
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Worst pain | 0-14 days
  NRS scale, 0-10
Average pain | 0-14 days
  NRS scale, 0-10

SECONDARY OUTCOMES:
analgesic methods | 0-14 days
  list of drugs (dose and duration) and other analgesic measures

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Anesthesiology, Oslo University Hospital, Ullevaal, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No